CLINICAL TRIAL: NCT05995275
Title: A Randomised, Placebo-Controlled, Dose-Ranging, Observer-Blind Phase 1/2 Study to Evaluate the Safety, Tolerability, and Immunogenicity of mRNA-1769 in Healthy Participants
Brief Title: A Study to Investigate The Safety, Tolerability, And Immune Response of a Range of Doses of mRNA-1769 Compared With Placebo in Healthy Participants From ≥18 Years of Age to <50 Years of Age
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: ModernaTX, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Prevention
Other Study IDs: mRNA-1769-P101
Record Dates: First submitted 2023-08-09; First posted 2023-08-16 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Smallpox; Mpox
Keywords: mRNA-1769 vaccine; mRNA-1769; Moderna
MeSH Terms: conditions — Smallpox; Mpox, Monkeypox

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- mRNA-1769 Dose A (Experimental): Participants will receive intramuscular (IM) injection of mRNA-1769 at Dose A on Day 1 and Day 29.
  Interventions: Biological: mRNA-1769
- mRNA-1769 Dose B (Experimental): Participants will receive IM injection of mRNA-1769 at Dose B on Day 1 and Day 29.
  Interventions: Biological: mRNA-1769
- mRNA-1769 Dose C (Experimental): Participants will receive IM injection of mRNA-1769 at Dose C on Day 1 and Day 29.
  Interventions: Biological: mRNA-1769
- Placebo (Placebo Comparator): Participants will receive IM injection of placebo matched to mRNA-1769 on Day 1 and Day 29.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: mRNA-1769 — Sterile liquid for injection
  Arms: mRNA-1769 Dose A; mRNA-1769 Dose B; mRNA-1769 Dose C
Other: Placebo — 0.9% sodium chloride injection (normal saline)
  Arms: Placebo

SUMMARY:
The goal of this study is to assess the safety, tolerability and immunogenicity of mRNA-1769 in healthy adult participants.

ELIGIBILITY:
Inclusion Criteria:

* Has a body mass index (BMI) between ≥18 kilogram per square meter (kg/m^2) to ≤39 kg/m^2.
* For female participants of childbearing potential: must have a negative highly sensitive pregnancy test with 28 days before the first dose of study drug, uses approved contraception during the study intervention period and for at least 3 months after the last dose of study drug, and not currently breastfeeding.

Exclusion Criteria:

* History of smallpox vaccination, vaccination with any poxvirus-based vaccine, history of of/or recent exposure to Mpox (MPX) (defined as close contact with a confirmed case of MPX within the past 14 days).
* Participant should not have any significant, progressive, unstable, or uncontrolled clinical condition, including any condition that may affect participant safety, assessment of safety endpoints, assessment of immune response, or adherence to study procedures per Investigator judgement.
* Participant is undergoing investigations for a potential chronic medical disorder.
* Bleeding disorder considered a contraindication to IM injection or phlebotomy.
* Dermatologic conditions that could affect local solicited AR assessments.
* History of anaphylactic reaction or allergic reactions that required medical intervention following any vaccine.
* Known or suspected allergy to any component of mRNA-1769.
* History of malignancy within previous 10 years (excluding non-melanoma skin cancer).
* Participant has any medical, psychiatric, or occupational condition, including reported history of drug or alcohol abuse, that, in the opinion of the Investigator, might pose additional risk due to participation in the study or could interfere with the interpretation of study results.
* Participant has received systemic immunosuppressants or immune-modifying drugs for >14 days in total within 6 months prior to Screening (for corticosteroids, ≥10 mg/day of prednisone or equivalent) or is anticipating the need for immunosuppressive treatment at any time during participation in the study. Topical tacrolimus is allowed if not used within 14 days prior to the day of enrolment. Participants may be rescheduled for enrolment if they no longer meet this criterion within the Screening Period. Inhaled, nasal, and topical steroids are allowed.
* Receipt or planned receipt of: Any vaccine(s), authorised or approved by local health agency, including mRNA vaccine, ≤28 days prior to the first injection through 28 days after the last dose of investigational (IMP).
* Intravenous blood products (red cells, platelets, immunoglobulins) within 3 months prior to the first injection up to the end of the study.
* Participated in an interventional study/received an investigational product within 28 days prior to the Screening Period or plans to do so while enroled in this study.

Note: Other inclusion and exclusion criteria may apply.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 351 (Actual)
Dates: Start 2023-08-15 (Actual); Primary Completion 2025-07-08 (Actual); Study Completion 2025-07-08 (Actual)

PRIMARY OUTCOMES:
Number of Solicited Local and Systemic Reactogenicity Adverse Reactions (ARs) Through 7 Days After Each Investigational Medicinal Product (IMP) | Up to Day 35
Number of Unsolicited Adverse Events (AEs) Through 7 Days After Each IMP | Up to Day 57
Number of Participants with Medically-Attended AEs (MAAEs) | Day 1 up to Day 395
Number of Participants with Adverse Events of Special Interest (AESIs) | Day 1 up to Day 395
Number of Participants with Serious Adverse Events (SAEs) | Day 1 up to Day 395
Number of Participants with AEs Leading to Study and/or Treatment Discontinuation | Day 1 up to Day 395

SECONDARY OUTCOMES:
Geometric Mean Titer (GMT) of Neutralising Antibody (nAb) against Mpox Virus (MPXV) by Plaque reduction neutralisation test (PRNT) | Days 1 and 43
Percentage of Participants With Seroconversion Based on Neutralising Antibody Responses Against MPXV | Days 1 and 43
Geometric Mean Concentration of Binding Antibodies (bAbs) Against MPXV Antigens by Meso Scale Discovery (MSD) Assay | Days 1, 29, 43, and 57
Percentage of Participants With Seroconversion Based on Binding Antibodies (bAb) Responses against MPXV | Days 1, 29, 43, and 57
Geometric Mean Titer of Neutralising Antibody Against Vaccinia Virus (VACV) by Plaque Reduction Neutralisation Test (PRNT) | Days 1 and 43
Percentage of Participants With Seroconversion Based on Neutralising Antibody Responses Against Vaccinia Virus | Days 1 and 43
Geometric Mean Concentration of Binding Antibodies Against Vaccinia Virus Antigens by Meso Scale Discovery Assay | Days 1, 29, 43, and 57
Percentage of Participants With Seroconversion Based on Binding Antibodies Responses Against Vaccinia Virus | Days 1, 29, 43, and 57

CONTACTS AND LOCATIONS:
Locations (12):
- United Kingdom (12):
  - Bradford Teaching Hospitals NHS Foundation Trust, Bradford
  - University Hospitals Bristol and Weston NHS Foundation Trust, Bristol
  - Lakeside Healthcare Research, Corby
  - University Hospitals of Leicester, Leicester
  - Liverpool University Hospitals NHS Foundation Trust, Liverpool
  - Barts Health NHS Trust, London
  - University College London Hospitals, London
  - Royal Free London NHS Foundation Trust, London
  - Chelsea and Westminster Hospital NHS Foundation Trust, London
  - Medicines Evaluation Unit, Manchester
  - Centre for Clinical Vaccinology and Tropical Medicine (CCVTM), Oxford
  - North Wales Clinical Research Facility Centre, Wrexham